CLINICAL TRIAL: NCT03730454
Title: A Multi-Center Randomized Trial of Transanastomotic Tube for Proximal Esophageal Atresia With Distal Tracheoesophageal Fistula Repair
Brief Title: Transanastomotic Tube for Proximal Esophageal Atresia With Distal Tracheoesophageal Fistula Repair
Acronym: TEF
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Phoenix Children's Hospital (Other)
Responsible Party: Principal Investigator, Justin Lee, MD, Pediatric Surgeon, Phoenix Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-136
Record Dates: First submitted 2018-11-01; First posted 2018-11-05 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Esophageal Atresia; Tracheoesophageal Fistula
MeSH Terms: conditions — Esophageal Atresia; Tracheoesophageal Fistula

STUDY DESIGN:
Intervention Model Description: Multisite randomized control trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Group A. Transanastomotic Tube (Experimental): Group A. Transanastomotic Tube: Standard repair of EA/TEF will be performed. TT will be used during the esophageal anastomosis creation.
  Interventions: Device: Transanastomotic Tube (5FR)
- Group B. No Transanastomotic Tube (Experimental): Group B. No Transanastomotic tube group: Standard repair of EA/TEF will be performed. TT will NOT be used during the esophageal anastomosis creation.
  Interventions: Other: No Transanastomotic Tube

INTERVENTIONS:
Device: Transanastomotic Tube (5FR) — 5FR tube left in place for 5 days after completion of esophageal anastomosis.
  Arms: Group A. Transanastomotic Tube
Other: No Transanastomotic Tube — No transanastomotic tube used during repair
  Arms: Group B. No Transanastomotic Tube

SUMMARY:
This trial will compare the effectiveness of two common surgical practices for Type C esophageal atresia repair: esophageal atresia (EA) with distal tracheoesophageal fistula (TEF). Infants with EA/TEF requiring surgical intervention will be recruited. Subjects will be randomized to either repair with or without transanstomotic tube (TT) during esophageal anastomosis creation. Primary outcome is symptomatic anastomotic stricture development requiring dilation within 12 months.

DETAILED DESCRIPTION:
Esophageal atresia is a congenital condition requiring surgical intervention. The most common configuration is Gross type C, proximal EA with distal TEF (EA/TEF). The operation for type C includes tracheoesophageal fistula closure and esophageal anastomosis creation. Although mortality has markedly decreased since the operation was first described, overall complication rate remains at 62%, with the most common complication being anastomotic stricture, 43%.

During the creation of esophageal anastomosis, two common practices are to either use or not use a transanastomtic tube (TT) across the anastomosis. However the utility and benefits of TT have not been validated. A recent retrospective analysis by the Midwestern Pediatric Surgical Research Consortium identified anastomotic stricture to be the most common postoperative complications (43%). On univariate analysis, only utilization of a TT was significantly associated with strictures (p=0.013). On multivariate analysis after adjusting for both pre and perioperative variables, TT use remained significant with an odd ratio (OR) of 1.91 (p=0.04).

Given the inherent limitations and biases of retrospective analysis, there is a critical need for a prospective multi-institutional study to validate this finding. The Western Pediatric Surgical Research Consortium (WPSRC) consists of 10 children's hospitals including Phoenix Children's Hospital, Doernbecher Children's Hospital, Primary Children's Hospital, Lucile Packard Children's Hospital, Seattle Children's Hospital, Colorado Children's Hospital, Children's Hospital of Los Angeles, Rady Children's Hospital, Benioff Children's Hospital, and Children's Medical Center Dallas. The WPSRC will conduct a prospective randomized control trial comparing the effects of TT use. Target enrollment is 150. One group of patients will receive TTs and another group of patients will not receive TTs. We hypothesize that the use of TT will result in increased anastomotic stricture formation. Primary outcome is symptomatic anastomotic stricture requiring dilation within 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Infants diagnosed with type C esophageal atresia: proximal esophageal atresia and distal tracheoesophageal fistula
* Primary repair of the esophageal atresia within the first six months of life
* Minimum follow up of 1 year (12 months)

Exclusion Criteria:

* Other types of esophageal atresia without esophageal anastomosis creation
* Major anomaly that influences likelihood of developing primary outcome or affects surgical treatment considerations

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 142 (Actual)
Dates: Start 2018-05-11 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Anastomotic stricture | 12 months
  Symptomatic anastomotic stricture requiring dilation

SECONDARY OUTCOMES:
Anastomotic Leak | 12 months
  Anastomotic leak seen radiographically or in the operating room
Recurrent Fistula | 12 months
  Recurrent fistula seen radiographically or in the operating room
Vocal cord injury | 12 months
  vocal cord injury seen radiographically or in the operating room
Unplanned return to OR | 12 months
  Any unplanned return to opearting room
Duration of perenteral nutrition | 12 months
  Days requrining TPN
Length of Stay | 12 months
  Length of stay during hospitalization for primary repair

CONTACTS AND LOCATIONS:
Overall Officials: Justin Lee, MD, Principal Investigator — Phoenix Children's Hospital
Locations (10):
- United States (10):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Children's Hospital Los Angeles, Los Angeles, California
  - Rady Children's Hospital, San Diego, California
  - Benioff Children's Hospital, San Francisco, California
  - Lucile Packard Children's Hospital, Stanford, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Doernbecher Children's Hospital, Portland, Oregon
  - Children's Medical Center, Dallas, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-19): https://cdn.clinicaltrials.gov/large-docs/54/NCT03730454/Prot_SAP_001.pdf